CLINICAL TRIAL: NCT01139801
Title: Cervical Ripening for Induction of Labor: Misoprostol Versus Oxytocin in Conjunction With Foley Balloon
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Aultman Health Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2009 ED
Record Dates: First submitted 2010-06-07; First posted 2010-06-09 (Estimated); Results first posted 2018-08-24 (Actual); Last update posted 2018-08-24 (Actual); Status verified 2018-08

CONDITIONS: Induction of Labor
Keywords: Cervical Ripening; Rate of Cesearean Section
MeSH Terms: interventions — Oxytocin; Misoprostol

ARMS (2):
- Oxytocin (Active Comparator): Foley balloon placement with intravenous low dose oxytocin administration starting 2 milliunits per minute.
  Interventions: Drug: Oxytocin
- Misoprostol (Experimental): Misoprostol, 25 mcg, is placed intravaginally into the posterior fornix of the vagina in conjunction with Foley balloon placement
  Interventions: Drug: Misoprostol

INTERVENTIONS:
Drug: Oxytocin — Foley balloon placement with intravenous low dose oxytocin administration starting 2 milliunits per minute.
  Other Names: pitocin
  Arms: Oxytocin
Drug: Misoprostol — Misoprostol, 25 mcg, is placed intravaginally into the posterior fornix of the vagina in conjunction with Foley balloon placement
  Other Names: cytotec
  Arms: Misoprostol

SUMMARY:
The purpose of this study is to specifically investigate the efficacy of an alternative pharmacologic cervical ripening agent, misoprostol, versus the standard oxytocin, as an adjunct to Foley balloon for induction of the unfavorable cervix.

DETAILED DESCRIPTION:
The design of this study is a randomized, controlled study with two arms. Both groups will undergo placement of a Foley catheter, through the external and internal os of the cervix, according to standard practice. In group A, receiving intravenous infusion of oxytocin, will serve as the control group as it is standard protocol at Aultman Hospital. Group B, intravaginal placement of misoprostol, will serve as the experimental group. The expected duration of participation begins at induction of labor and concludes at time of delivery.

ELIGIBILITY:
Inclusion Criteria:

* Participant or surrogate is capable of giving informed consent
* Anticipated number - 50 patients with 25 in each study arm Female with singleton gestation, live intrauterine pregnancy
* Participant is undergoing an indicated induction of labor
* Participant is found to have cervical Bishop score ≤5 on initial cervical exam
* Participant has no medical or obstetrical contraindications to induction of labor

Exclusion Criteria:

* Participant has ≥2 painful contractions in 10 min in 2 subsequent 10 min periods
* Manufacturer's contraindications to misoprostol or oxytocin

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2009-09; Primary Completion 2010-03 (Actual); Study Completion 2010-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Erica Downey, MD, Principal Investigator — Aultman Health Foundation
Locations (1):
- Aultman Health Foundation, Canton, Ohio, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Oxytocin | Misoprostol
Started | 25 | 25
Completed | 25 | 25
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Oxytocin | Misoprostol | Total
Number analyzed (Participants) | 25 | 25 | 50
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 25 | 25 | 50
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 25 | 25 | 50
  Male | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Rate of Induction To Delivery
Description: To assess effectiveness of misoprostol used in conjunction with Foley balloon versus the standard oxytocin regimen in regards to induction times
Time Frame: 24 hrs
Population: Patients requiring caesarean section excluded from analysis.
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Oxytocin | Misoprostol
Number analyzed (Participants) | 16 | 17
minutes | 732.19 (236.99) | 944.35 (317.78)
Statistical Analysis 1: Comparison: Oxytocin vs Misoprostol; Test type: Superiority; p = 0.037, t-test, 2 sided; Mean Difference (Final Values) = 212.2, 95% CI 2-sided [13.3 to 411.0]

2. Secondary Outcome: Delivery Route
Description: To assess for differences in delivery routes
Time Frame: 24 hrs
Measure: Count of Participants; unit: Participants
Arm/Group | Oxytocin | Misoprostol
Number analyzed (Participants) | 25 | 25
Participants
  Vagnial Delivery | 16 | 17
  Cesearean | 9 | 8

ADVERSE EVENTS:
Time Frame: 24 hours
Arm/Group | Oxytocin | Misoprostol
All-Cause Mortality (participants affected / at risk) | 0/25 | 0/25
Serious Adverse Events (participants affected / at risk) | 0/25 | 0/25
Other Adverse Events (participants affected / at risk) | 0/25 | 0/25

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No